CLINICAL TRIAL: NCT06793787
Title: Risk Evaluation by Coronary Imaging and Artificial Intelligence-Based Functional Analyzing Techniques: Plasma Proteomic Profiles of Atheroma Classified by Intracoronary Imaging.
Brief Title: Risk Evaluation by COronary Imaging and Artificial intelliGence Based fuNctIonal analyZing tEchniques - IV
Acronym: RECOGNIZE-IV
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, Director of Cardiology, Director of cardiovascular catherization lab, Principle Investigator Affiliation: Ruijin Hospital, Ruijin Hospital
Other Study IDs: 2022YFC2533502-4
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Coronary Atheroscleroses; Acute Coronary Syndromes (ACS); Chronic Coronary Syndrome
Keywords: Acute coronary syndrome; Chronic coronary syndrome; Coronary vulnerable plaque; intracoronary imaging; coronary CT angiography
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood samples collected at the same time of the coronary imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cornary plaque analysis group: Patients with CCS or NSTE-ACS, who have marginal or obstructive lesions (DS 40% - 90%) detected by CCTA or ICA, will be consecutively enrolled. OCT, with or without other intracoronary imaging modalities including IVUS and NIRS, will be performed to classify plaque types and precisely measure plaque burden and other geometric parameters. Plasma samples will be collected on the day of angiography in all patients after overnight fasting.

SUMMARY:
This study is a single-center, prospective cohort study. The study is designed to identify novel circulating biomarkers for early prediction of high-risk coronary plaques. Patients diagnosed with chronic coronary syndrome (CCS) or non-ST-segment elevation acute coronary syndrome (NSTE-ACS), with marginal lesions or obstructive lesions in major coronary arteries detected by noninvasive coronary CT angiography (CCTA) or invasive coronary angiography (ICA), will be consecutively enrolled. Optical coherence tomography (OCT), with or without other intracoronary imaging modalities such as intravascular ultrasound (IVUS) and near infrared spectroscopy (NIRS), will be performed. Liquid chromatography-mass spectrometry (LC-MS/MS), bioinformatic analysis, and machine learning methods will be performed to characterize plasma proteomic profiles. The cohort will be followed-up every 3 months for 2 years. The association of novel biomarkers with the occurrence of major adverse cardiovascular events (MACEs) will be examined.

DETAILED DESCRIPTION:
This study is a single-center, prospective cohort study. The study is designed to identify novel circulating biomarkers for early prediction of high-risk plaques. Patients diagnosed with chronic coronary syndrome (CCS) or non-ST-segment elevation acute coronary syndrome (NSTE-ACS), with marginal lesions (diameter stenosis [DS] between 40%-69%) or obstructive lesions (DS ≥70% or CT-FFR/FFR <0.8) in major coronary arteries detected by noninvasive coronary CT angiography (CCTA) or invasive coronary angiography (ICA), will be consecutively enrolled. Optical coherence tomography (OCT), with or without other intracoronary imaging modalities including intravascular ultrasound (IVUS) and near infrared spectroscopy (NIRS), will be performed to precisely measure plaque burden and other geometric parameters.

Under the guidance of OCT, these plaques will be classified into different types (intimal xanthoma, early and late fibroatheroma, thin-cap fibroatheroma [TCFA], plaque rupture [PR], plaque erosion [PE], calcified nodules, healed lesions). If IVUS is additionally performed, total atheroma volume (TAV), percent atheroma volume (PAV), and remodeling index will be calculated. If NIRS is additionally performed, lipid core burden index (LCBI) will be calculated. Integrated analysis will also be performed to investigate the relationship between plaque characteristics obtained from different imaging modalities.

Afterwards, liquid chromatography-mass spectrometry (LC-MS/MS), bioinformatic analysis, and machine learning methods will be performed to characterize plasma proteomic profiles in patients with different types of coronary atherosclerotic plaques. Differentially expressed proteins will be analyzed to identify novel biomarkers for high-risk plaques.

The cohort will be followed-up every 3 months for 2 years. The association of novel biomarkers with the occurrence of major adverse cardiovascular events (MACEs) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with CCS or NSTE-ACS
* Receive CCTA scan or ICA, with marginal lesions (DS between 40%-69%) or obstructive lesions (DS ≥70% or CT-FFR/FFR <0.8) in major coronary arteries
* Receive invasive coronary angiography and OCT, with or without other intracoronary imaging techniques such as IVUS and NIRS

Exclusion Criteria:

* Receive percutaneous coronary intervention (PCI) within 6 months
* Prior history of myocardial infarction or heart failure
* Prior history of coronary artery bypass graft (CABG)
* Abnormal liver function (serum alanine aminotransferase [ALT] level exceeding 3 times the upper limit of normal) or abnormal kidney function (eGFR ≤30%)
* Familial hypercholesterolemia
* Estimated survival ≤ 1 year
* Malignant tumor
* Pregnant or lactation, or have the intention to give birth within one year
* Poor compliance, unable to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with chronic coronary syndrome (CCS) or non-ST-segment elevation acute coronary syndrome (NSTE-ACS), with marginal lesions (diameter stenosis [DS] between 40%-69%) or obstructive lesions (DS ≥70% or CT-FFR/FFR <0.8) in major coronary arteries detected by noninvasive coronary CT angiography (CCTA) or invasive coronary angiography (ICA), will be consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction performance of high-risk plaques by novel biomarkers | 2 years
  The prediction performance of high-risk plaques (area under receiver operating characteristics curve, etc.) by novel biomarkers will be compared with traditional risk factors.

SECONDARY OUTCOMES:
Major cardiovascular events (MACEs) | 2 years
  A composite endpoint of cardiovascular death, non-fatal myocardial infarction, and unplanned revascularization during follow-up. The prediction performance of MACEs by novel biomarkers and traditional risk factors will be compared.
Cardiovascular death | 2 years
  The occurrence of cardiovascular death during follow-up. The prediction performance of cardiovascular death by novel biomarkers and traditional risk factors will be compared.
Myocardial infarction | 2 years
  The occurrence of myocardial infarction during follow-up. The prediction performance of myocardial infarction by novel biomarkers and traditional risk factors will be compared.
Unplanned revascularization | 2 years
  The occurrence of unplanned revascularization during follow-up. The prediction performance of novel biomarkers and traditional risk factors will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D.,Ph.D., Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided